CLINICAL TRIAL: NCT01305733
Title: Local Infiltration Analgesia During Total Knee Arthroplasty - Reduced Opiate Consumption and Faster Mobilisation Postoperatively - Randomized Controlled Trial
Brief Title: Local Infiltration Analgesia During Total Knee Arthroplasty
Acronym: LIA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Coxa, Hospital for Joint Replacement (Other)
Responsible Party: Principal Investigator, Mika Niemeläinen, orthopaedic surgeon, Coxa, Hospital for Joint Replacement
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Coxa - LIA
Record Dates: First submitted 2011-02-28; First posted 2011-03-01 (Estimated); Last update posted 2012-05-09 (Estimated); Status verified 2012-05

CONDITIONS: Pain
Keywords: Pain relief
MeSH Terms: conditions — Pain | interventions — Ketorolac; Epinephrine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- local infiltration analgesia (Active Comparator): The injectant mixture consists of 150 mg levobupivacaine mixed with 30 mg ketorolac and 0.5 mg adrenaline
  Interventions: Drug: The injectant mixture consists of 150 mg levobupivacaine mixed with 30 mg ketorolac and 0.5 mg adrenaline
- saline injection (Placebo Comparator): The normal saline injection are used in the control group in the same manner than in the RKA group.
  Interventions: Other: saline injection

INTERVENTIONS:
Drug: The injectant mixture consists of 150 mg levobupivacaine mixed with 30 mg ketorolac and 0.5 mg adrenaline — The injectant mixture consists of 150 mg levobupivacaine mixed with 30 mg ketorolac and 0.5 mg adrenaline
  Arms: local infiltration analgesia
Other: saline injection — saline
  Arms: saline injection

SUMMARY:
The primary objective is to evaluate whether local infiltration analgesia (LIA) will reduce oxycodone consumption during the first 48 postoperative hours in patients undergoing total knee arthroplasty (TKA).

DETAILED DESCRIPTION:
The goal of LIA is to gain an effective and safe pain control during the first postoperative days. The study is a single-center, randomized controlled trial, which will be performed in Coxa Hospital for Joint Replacement in Tampere, Finland. The injectant mixture consists of 150 mg levobupivacaine mixed with 30 mg ketorolac and 0.5 mg adrenaline with occasional variations if the patient is unusually small, very elderly, infirm or has a history of significant intolerance to analgesics or anesthetic agents. The RKA mixture is diluted with normal saline. Total volume of the solution is 100 ml depending on the size of the wound. The normal saline injection are used in the control group in the same manner than in the RKA group.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring primary TKA for primary OA
* Patients aged 75 years or less
* Patients suitable for all applicable devices

Exclusion Criteria:

* Rheumatoid arthritis or other inflammatory diseases
* Patients requiring bone grafting during surgery
* Unwilling to provide informed consent
* BMI > 35
* ASA > 3
* Renal dysfunction
* Allergic to ASA
* Previous high tibial osteotomy or previous osteosynthesis
* > 15 degrees varus / valgus malalignment
* Physical, emotional or neurological conditions which would comprise the patient´s compliance with postoperative rehabilitation and follow-up (e.g. drug or alcohol abuse, serious mental illness, general neurological conditions such as Parkinson, MS, etc.)
* Known sensitivity to materials in the devices

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-03; Primary Completion 2012-05 (Actual); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
oxycodone consumption during the first 48 postoperative hours | 48 hours

SECONDARY OUTCOMES:
functional outcome after TKA | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Antti Eskelinen, M.D., Ph.D, Study Director — Coxa, Hospital for Joint Replacement; Mika Niemeläinen, MD, Principal Investigator — Coxa, Hospital for Joint Replacement
Locations (2):
- Finland (2):
  - Coxa - hospital for joint replacement, Tampere, Pirkanmaa
  - COXA, Tampere, Pirkanmaa